CLINICAL TRIAL: NCT05531617
Title: A Prospective,Randomised, Open Label Study for Comparison of the Incidence and Severity of Postoperative Sore Throat (POST) Using C-MAC Video Laryngoscope and Traditional Macintosh Laryngoscope for Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seth Gordhandas Sunderdas Medical College (Other)
Responsible Party: Principal Investigator, Gousmahammad Myageri, Senior Resident, Seth Gordhandas Sunderdas Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: EC/202/2018
Record Dates: First submitted 2022-09-01; First posted 2022-09-08 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Hoarseness of Voice; Sore-throat
Keywords: Endotracheal tube; Postoperative sore throat; Hoarseness of voice; Macintosh laryngoscope; C-MAC video laryngoscope
MeSH Terms: conditions — Hoarseness; Pharyngitis | interventions — Intubation

STUDY DESIGN:
Intervention Model Description: A prospective,randomised, open label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- M group (Active Comparator): Group Intubated with Macintosh laryngoscope is labelled as M group
  Interventions: Procedure: Intubation
- V group (Active Comparator): Group Intubated with C-Mac video laryngoscope is labelled as V group
  Interventions: Procedure: Intubation

INTERVENTIONS:
Procedure: Intubation — Study groups Intubated with Macintosh or cmac video laryngoscopes

SUMMARY:
The aim of this study is to compare the incidence of postoperative sore throat after intubation with two different types of laryngoscopes.

DETAILED DESCRIPTION:
Postoperative sore throat is a well known complication after endotracheal intubation. One of the major contributing factors is trauma associated with laryngoscopy. With decreased force applied to visualise cords, video laryngoscopes should decrease the incidence of postoperative sore throat. In this study we compared the incidence and severity of postoperative sore throat when laryngoscopy was done using c-mac video laryngoscope D-blade( group V) versus Macintosh laryngoscope (Group M). Method: Fifty four American society of Anaesthesiologists (ASA) 1&2 patients between age 18-60 years , undergoing laproscopic surgeries of short duration were included in this study and laryngoscopy was done with Macintosh laryngoscope in M group and with C MAC video laryngoscope D blade in V group. Patients were followed up 2hours, 6hours, 12hours and 24hours in postoperative period to see postoperative sore throat and hoarseness of voice .

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 years
* American society of Anaesthesiologists(ASA)1 and 2
* Mallampati (MPC) grading 1 and 2
* laparoscopic cholecystectomy and appendectomy
* Surgeries of short duration(<2hour)

Exclusion Criteria:

* Patients refusing to give consent
* Pregnant and lactating patients
* Patients with severe co-morbidities requiring postoperative ventilatory support

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
The incidence and severity of postoperative sore throat measured | Upto 24 hours after surgery
  The incidence and severity of Postoperative sore throat is measured after surgery at 2hours, 6hours, 12hours and 24 hours based on a scaling system as described below
  * No sore throat at any time since the operation Grade 0
  * Minimal - patient answered in the affirmative when asked about sore throat - Grade1
  * Moderate - patient complained of sore throat on his/her own - Grade 2
  * Severe - patient is in obvious distress-Grade 3

SECONDARY OUTCOMES:
The incidence and severity of Hoarseness of voice | Upto 24 hours after surgery
  The incidence and severity of Postoperative hoarseness of voice measured at 2hours, 6hours, 12hours and 24hours post surgery by scaling system as described below
  * No complaint of hoarseness at any time since the operation - Grade 0
  * Minimal - minimal change in quality of speech. Patient answers in the affirmative only when enquired about - Grade 1
  * Moderate - moderate change in quality of speech of which the patient complains on his/her own - Grade 2
  * Severe - gross change in the quality of voice perceived by the observer - Grade 3

CONTACTS AND LOCATIONS:
Locations (1):
- Seth GSMC and KEM Hospital, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tosh P, Kadapamannil D, Rajan S, Narayani N, Kumar L. Effect of C-MAC Video Laryngoscope-aided intubations Using D-Blade on Incidence and Severity of Postoperative Sore Throat. Anesth Essays Res. 2018 Jan-Mar;12(1):140-144. doi: 10.4103/aer.AER_182_17. PMID 29628570
- [Background] Aqil M, Khan MU, Mansoor S, Mansoor S, Khokhar RS, Narejo AS. Incidence and severity of postoperative sore throat: a randomized comparison of Glidescope with Macintosh laryngoscope. BMC Anesthesiol. 2017 Sep 12;17(1):127. doi: 10.1186/s12871-017-0421-4. PMID 28899338